CLINICAL TRIAL: NCT00776425
Title: Quality of Life Related Response to Treatment in Anemic Cancer Patients Receiving Recormon and Efficacy of the Drug Dosage 30,000 IU Once Weekly in Patients With Lymphoproliferative Disorders
Brief Title: A Study of the Quality of Life and Treatment Response to Once Weekly Epoetin Beta (Recormon) Treatment in Anemic Participants With Solid and Lymphoid Malignancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20197
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (2):
- Epoetin Beta 150 IU/kg (Experimental): Participants with solid and lymphoid malignancies will receive subcutaneous or intravenous epoetin beta at a dose of 150 IU per kg of body weight thrice weekly.
  Interventions: Drug: Epoetin beta
- Epoetin Beta 30000 IU (Experimental): Participants with lymphoid malignancies will receive subcutaneous or intravenous epoetin beta at a dose of 30000 IU once weekly.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Epoetin beta subcutaneously or intravenously at a dose of 150 IU per kg of body weight thrice weekly or 30000 IU once weekly.
  Other Names: Recormon

SUMMARY:
This 2 arm study will investigate Quality of Life response in anemic participants with solid and lymphoid malignancies, who are receiving concomitant chemotherapy. Participants with solid and lymphoid malignancies will receive epoetin beta at a dose of 150 international units per kilogram (IU/kg) three times weekly. Participants with lymphoid malignancies will receive epoetin beta 30000 IU once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Anemia and prescribed treatment with epoetin beta
* Confirmed diagnosis of a solid or lymphoid hematologic malignancy
* Receiving or scheduled to receive chemotherapy
* Life expectancy of greater than or equal to (>=6) months

Exclusion Criteria:

* Anemia after bleeding, hemolytic anemia, megaloblastic anemia, anemia in chronic kidney failure, lever and endocrinology diseases
* Contraindications to epoetin beta
* Administration of epoetin beta during chemotherapy (e.g., on the third day after chemotherapy cycle start)
* Bleeding within one month before and/or during study
* Severe infection within one month before and/or during study
* Inability of participant to fill the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved a Clinical Response 3-4 Weeks After Start of Treatment | 3-4 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by greater than or equal to (>=) 2 grams per liter (g/L) against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received 150 IU/kg and those received 30000 IU doses.
Percentage of Participants Who Achieved a Clinical Response 6-8 Weeks After Start of Treatment | 6-8 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received 150 IU/kg and those received 30000 IU doses.
Percentage of Participants Who Achieved a Clinical Response 10-12 Weeks After Start of Treatment | 10-12 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received 150 IU/kg and those received 30000 IU doses.
Percentage of Participants Who Achieved a Clinical Response 3-4 Weeks After Start of Treatment with Mixed Dosing Regimen | 3-4 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Percentage of Participants Who Achieved a Clinical Response 6-8 Weeks After Start of Treatment with Mixed Dosing Regimen | 6-8 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Percentage of Participants Who Achieved a Clinical Response 10-12 Weeks After Start of Treatment with Mixed Dosing Regimen | 10-12 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants who received initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Quality of Life of Anemic Participants Using Short Form 36 (SF-36) Questionnaire Prior To Treatment | Baseline
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants.
Quality of Life of Anemic Participants Using SF-36 Questionnaire 3-4 Weeks After Start of Treatment | 3-4 Weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants.
Quality of Life of Anemic Participants Using SF-36 Questionnaire 6-8 Weeks After Start of Treatment | 6-8 Weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants.
Quality of Life of Anemic Participants Using SF-36 Questionnaire 10-12 Weeks After Start of Treatment | 10-12 Weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants.
Percentage of Participants With Quality of Life Integral Value (IV) Reduction Prior To Treatment | Baseline
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a population norm (nIV). The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Percentage of Participant With Quality of Life IV Reduction 3-4 Weeks After Start of Treatment | 3-4 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Percentage of Participant With Quality of Life IV Reduction 6-8 Weeks After Start of Treatment | 6-8 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Percentage of Participant With Quality of Life IV Reduction 10-12 Weeks After Start of Treatment | 10-12 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Percentage of Participant With Characteristics of The Quality of Life Related Response To Treatment 3-4 Weeks After Start of Treatment | 3-4 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization.
Percentage of Participant With Characteristics of The Quality of Life Related Response To Treatment 6-8 Weeks After Start of Treatment | 6-8 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization.
Percentage of Participant With Characteristics of The Quality of Life Related Response To Treatment 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization.
Fatigue Severity Score at Baseline | Baseline
  Fatigue was assessed by a digital rating scale (0 to 10) of MD Anderson Symptom Inventory (MDASI) cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Fatigue Severity Score 3-4 Weeks After Start of Treatment | 3-4 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Fatigue Severity Score 6-8 Weeks After Start of Treatment | 6-8 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Fatigue Severity Score 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participant With Various Fatigue Severity Prior To Treatment | Baseline
  Fatigue was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participant With Various Fatigue Severity 3-4 Weeks After Start of Treatment | 3-4 Weeks
  Fatigue was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participant With Various Fatigue Severity 6-8 Weeks After Start of Treatment | 6-8 Weeks
  Fatigue was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participant With Various Fatigue Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Fatigue was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participant With Different Symptoms Prior to Treatment (MDASI Questionnaire) | Baseline
  Percentage of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented.
Percentage of Participant With Different Symptoms 3-4 Weeks After Start of Treatment (MDASI Questionnaire) | 3-4 Weeks
  Percentage of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented.
Percentage of Participant With Different Symptoms 6-8 Weeks After Start of Treatment (MDASI Questionnaire) | 6-8 Weeks
  Percentage of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented.
Percentage of Participant With Different Symptoms 10-12 Weeks After Start of Treatment (MDASI Questionnaire) | 10-12 Weeks
  Percentage of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented.
Severity Score of Different Symptoms Prior toTreatment (MDASI Questionnaire) | Baseline
  Symptoms' type was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. Severity grades used for assessment of symptoms severity: 1) Minor symptom, score 1-4; 2) Moderate symptom: score 5-6 and Severe symptom: Score 7-10).
Severity Score of Different Symptoms 3-4 Weeks After Start of Treatment (MDASI Questionnaire) | 3-4 weeks
  Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following severity grades were used for assessment of symptoms severity: 1) minor symptom, score 1-4; 2) moderate symptom: score 5-6; and 3) severe symptom: score 7-10.
Severity Score of Different Symptoms 6-8 Weeks After Start of Treatment (MDASI Questionnaire) | 6-8 Weeks
  Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following severity grades were used for assessment of symptoms severity: 1) minor symptom, score 1-4; 2) moderate symptom: score 5-6; and 3) severe symptom: score 7-10.
Severity Score of Different Symptoms 10-12 Weeks After Start of Treatment (MDASI Questionnaire) | 10-12 Weeks
  Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following severity grades were used for assessment of symptoms severity: 1) minor symptom, score 1-4; 2) moderate symptom: score 5-6; and 3) severe symptom: score 7-10.
Percentage of Participants With Improvement in Symptoms Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Symptoms' type was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. Severity grades used for assessment of symptoms severity: 1) Minor symptom, score 1-4; 2) Moderate symptom: score 5-6 and Severe symptom: Score 7-10).
Percentage of Participants With Concomitant Symptoms of Various Severity Prior To Treatment | Baseline
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms; 3) Only mild symptoms (score 1-4).
Percentage of Participants With Concomitant Symptoms of Various Severity 3-4 Weeks After Start of Treatment | 3-4 weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms; 3) Only mild symptoms (score 1-4).
Percentage of Participants With Concomitant Symptoms of Various Severity 4-6 Weeks After Start of Treatment | 4-6 weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms; 3) Only mild symptoms (score 1-4).
Percentage of Participants With Concomitant Symptoms of Various Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms; 3) Only mild symptoms (score 1-4).
Quality of Life of Anemic Participants With Clinical Response Using SF-36 Questionnaire Prior To Treatment | Baseline
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Quality of Life of Anemic Participants With Clinical Response Using SF-36 Questionnaire 3-4 Weeks After Start of Treatment | 3-4 weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Quality of Life of Anemic Participants With Clinical Response Using SF-36 Questionnaire 6-8 Weeks After Start of Treatment | 6-8 weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Quality of Life of Anemic Participants With Clinical Response Using SF-36 Questionnaire 10-12 Weeks After Start of Treatment | 10-12 weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Percentage of Participants With Different Symptoms Who Had Clinical Response Prior to Treatment | Baseline
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L with no blood transfusions within the 6 previous weeks.
Percentage of Participants With Different Symptoms Who Had Clinical Response 3-4 Weeks After Start of Treatment | 3-4 weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Percentage of Participants With Different Symptoms Who Had Clinical Response 6-8 Weeks After Start of Treatment | 6-8 weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Percentage of Participants With Different Symptoms Who Had Clinical Response 10-12 Weeks After Start of Treatment | 10-12 weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Severity Score of Different Symptoms in Anemic Participants With Clinical Response Prior To Treatment | Baseline
  Severity grades on a scale of 0-10, were used for assessment of symptoms severity: 1) Minor symptom, score 1-4; 2) Moderate symptom: score 5-6 and Severe symptom: Score 7-10). Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Severity Score of Different Symptoms in Anemic Participants With Clinical Response 3-4 Weeks After Start of Treatment | 3-4 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Severity Score of Different Symptoms in Anemic Participants With Clinical Response 6-8 Weeks After Start of Treatment | 6-8 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Severity Score of Different Symptoms in Anemic Participants With Clinical Response 10-12 Weeks After Start of Treatment | 10-12 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >=2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Percentage of Participants With Clinical Response After First 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 3-4 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Percentage of Participants With Clinical Response After Second 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 6-8 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Percentage of Participants With Clinical Response After Third 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 10-12 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results were presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Quality of Life in Anemic Participants Receiving Treatment at 30000 IU Once Weekly (SF-36 Questionnaire) Prior to Treatment | Baseline
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Quality of Life in Anemic Participants Receiving Treatment at 30000 IU Once Weekly (SF-36 Questionnaire) 3-4 Weeks After Start of Treatment | 3-4 weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Quality of Life in Anemic Participants Receiving Treatment at 30000 IU Once Weekly (SF-36 Questionnaire) 6-8 Weeks After Start of Treatment | 6-8 Weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Quality of Life in Anemic Participants Receiving Treatment at 30000 IU Once Weekly (SF-36 Questionnaire) 10-12 Weeks After Start of Treatment | 10-12 Weeks
  The SF-36 evaluates 36 questions related to participant-rated quality of life using 7 domains: physical and social functioning, physical and emotional role limitations, overall health, vitality, and mental health. The total score is the average of the individual question scores, which is scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Lymphoproliferative Disorders and Solid Tumors Who Had Quality of Life IV Reduction Prior to Treatment | Baseline
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minimal reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Severe reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV). Results are presented for participants with lymphoproliferative disorders and solid tumors.
Number of Participants With Lymphoproliferative Disorders and Solid Tumors Who Had Quality of Life IV Reduction 3-4 Weeks After Start of Treatment | 3-4 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minimal reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Severe reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV). Results are presented for participants with lymphoproliferative disorders and solid tumors.
Number of Participants With Lymphoproliferative Disorders and Solid Tumors Who Had Quality of Life IV Reduction 6-8 Weeks After Start of Treatment | 6-8 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minimal reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Severe reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV). Results are presented for participants with lymphoproliferative disorders and solid tumors.
Number of Participants With Lymphoproliferative Disorders and Solid Tumors Who Had Quality of Life IV Reduction 10-12 Weeks After Start of Treatment | 10-12 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minimal reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Severe reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV). Results are presented for participants with lymphoproliferative disorders and solid tumors.
Percentage of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors Prior Receiving Treatment at 30000 IU Once Weekly | Baseline
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results were presented for participants with lymphoproliferative disorders (LD) and solid tumors (STS) who received 30000 IU dose.
Percentage of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 3-4 Weeks After Start of Treatment at 30000 IU Once Weekly | 3-4 weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results were presented for participants with lymphoproliferative disorders (LD) and solid tumors (STS) who received 30000 IU dose.
Percentage of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 6-8 Weeks After Start of Treatment at 30000 IU Once Weekly | 6-8 weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results were presented for participants with lymphoproliferative disorders (LD) and solid tumors (STS) who received 30000 IU dose.
Percentage of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 10-12 Weeks After Start of Treatment at 30000 IU Once Weekly | 10-12 Weeks
  Percentage of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results were presented for participants with lymphoproliferative disorders (LD) and solid tumors (STS) who received 30000 IU dose.
Severity Score of Different Symptoms in Participants With Lymphoproliferative Disorders and Solid Tumors Prior to Treatment at 30000 IU Once Weekly | Baseline
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Severity Score of Different Symptoms in Participants With Lymphoproliferative Disorders and Solid Tumors 3-4 Weeks After Start of Treatment at 30000 IU Once Weekly | 3-4 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Severity Score of Different Symptoms in Participants With Lymphoproliferative Disorders and Solid Tumors 6-8 Weeks After Start of Treatment at 30000 IU Once Weekly | 6-8 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Severity Score of Different Symptoms in Participants With Lymphoproliferative Disorders and Solid Tumors 10-12 Weeks After Start of Treatment at 30000 IU Once Weekly | 10-12 weeks
  Severity grades on a scale of 0-10 were used for assessment of symptoms severity. The following severity grades were used: 1) Minor symptom: score 1-4; 2) Moderate symptom: score 5-6; and 3) Severe symptom: score 7-10. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Percentage of Participants With Improvement in Symptoms Severity Categorized by Lymphoproliferative Disorders and Solid Tumors 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Severity grades on a scale of 0-10, were used for assessment of symptoms severity: 1) Minor symptom, score 1-4; 2) Moderate symptom: score 5-6 and 3) Severe symptom: Score 7-10. Results were presented for participants with lymphoproliferative disorders (LD) and solid tumors (STS) who received 30000 IU dose.
Number of Participants Who Achieved a Clinical Response 3-4 Weeks After Start of Treatment | 3-4 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by greater than or equal to (>=) 2 grams per liter (g/L) against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received 150 IU/kg and those received 30000 IU doses.
Number of Participants Who Achieved a Clinical Response 6-8 Weeks After Start of Treatment | 6-8 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received 150 IU/kg and those received 30000 IU doses.
Number of Participants Who Achieved a Clinical Response 10-12 Weeks After Start of Treatment | 10-12 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received 150 IU/kg and those received 30000 IU doses.
Number of Participants Who Achieved a Clinical Response With Mixed Drug Dosing Regimen, 3-4 Weeks After Start of Treatment | 3-4 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Number of Participants Who Achieved a Clinical Response With Mixed Drug Dosing Regimen, 6-8 Weeks After Start of Treatment | 6-8 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received mixed dosing regimen with initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Number of Participants Who Achieved a Clinical Response With Mixed Dosing Regimen, 10-12 Weeks After Start of Treatment | 10-12 weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants who received mixed dosing regimen with initial dose at 150 IU/kg and those received initial dose at 30000 IU/kg doses.
Number of Participants With Quality of Life IV Reduction 3-4 Weeks After Start of Treatment | 3-4 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Number of Participants With Quality of Life IV Reduction 6-8 Weeks After Start of Treatment | 6-8 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Number of Participants With Quality of Life IV Reduction 10-12 Weeks After Start of Treatment | 10-12 Weeks
  A scale of the quality of life IV was developed for stratification of participants depending on the degree of lowering of the quality of life. The analysis has been performed based on the quality of life IV of a participant with a nIV. The following grades of the quality of life IV reduction were determined: 1) No quality of life reduction (no differences between participant IV and nIV); 2) Minor reduction of the IV quality of life (IV reduction at <25% of nIV); 3) Moderate reduction of the IV quality of life (IV reduction at 25-50% of nIV); 4) Significant reduction of the IV quality of life (IV reduction at 51-75% of nIV); 5) Critical reduction of the IV quality of life (IV reduction at >75% of nIV).
Number of Participants With Characteristics of the Quality of Life Related Response To Treatment 3-4 Weeks After Start of Treatment | 3-4 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization. Quality of life related responses to treatment was characterized as stabilization if no changes in the quality of life IV were observed. Quality of life related responses to treatment was characterized as improvement when quality of life IV was changed positively (positive changes in the quality of life IV).
Number of Participants With Characteristics of the Quality of Life Related Response To Treatment 6-8 Weeks After Start of Treatment | 6-8 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization. Quality of life related responses to treatment was characterized as stabilization if no changes in the quality of life IV were observed. Quality of life related responses to treatment was characterized as improvement when quality of life IV was changed positively (positive changes in the quality of life IV).
Number of Participants With Characteristics of the Quality of Life Related Response To Treatment 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Quality of life related response to treatment was determined for each participant. Depending on the change of grade of the quality of life IV, quality of life related responses to treatment were characterized as improvement or stabilization. Quality of life related responses to treatment was characterized as stabilization if no changes in the quality of life IV were observed. Quality of life related responses to treatment was characterized as improvement when quality of life IV was changed positively (positive changes in the quality of life IV).
Percentage of Participants With Various Fatigue Severity 3-4 Weeks After Start of Treatment | 3-4 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participants With Various Fatigue Severity 6-8 Weeks After Start of Treatment | 6-8 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Percentage of Participants With Various Fatigue Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Fatigue severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following fatigue grades were used: 1) Mild fatigue: score 1-3; 2) Moderate fatigue: score 4-6; 3) Severe fatigue: score 7-10. Score 1-3 fatigue was classified as insignificant; score 4-10 fatigue was assessed as significant.
Number of Participants With Different Symptoms 3-4 Weeks After Start of Treatment (MDASI Questionnaire) | 3-4 Weeks
  Number of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented. Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. Participants were asked to rate severity of each symptom; each item rated from 0 to 10, with 0 = symptom not present and 10 = severe symptom.
Number of Participant With Different Symptoms 6-8 Weeks After Start of Treatment (MDASI Questionnaire) | 6-8 Weeks
  Number of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented. Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. Participants were asked to rate severity of each symptom; each item rated from 0 to 10, with 0 = symptom not present and 10 = severe symptom.
Number of Participants With Different Symptoms 10-12 Weeks After Start of Treatment (MDASI Questionnaire) | 10-12 Weeks
  Number of participants with different symptoms (sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) of MDASI cancer participant symptom assessment questionnaire is presented. Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. Participants were asked to rate severity of each symptom; each item rated from 0 to 10, with 0 = symptom not present and 10 = severe symptom.
Number of Participants With Improvement in Symptoms Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following severity grades were used for assessment of symptoms severity: 1) minor symptom: score 1-4; 2) moderate symptom: score 5-6; and 3) severe symptom: score 7-10. Participants who had a reduction in scores from moderate-to-severe to mild were considered improved.
Number of Participants With Concomitant Symptoms of Various Severity 3-4 Weeks After Start of Treatment | 3-4 weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms (score >=5); 3) Only mild symptoms (score 1-4).
Number of Participants With Concomitant Symptoms of Various Severity 6-8 Weeks After Start of Treatment | 6-8 weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms (score >=5); 3) Only mild symptoms (score 1-4).
Number of Participants With Concomitant Symptoms of Various Severity 10-12 Weeks After Start of Treatment | 10-12 Weeks
  The number of concomitant symptoms was assessed in each participant. As a participant may concomitantly experience symptoms of various intensity, the following groups of participants were assessed based on the number and severity of symptoms: 1) >=7 moderate and severe symptoms (score >=5); 2) <7 moderate and severe symptoms (score >=5); 3) only mild symptoms (score 1-4).
Number of Participants With Different Symptoms Who Had Clinical Response 3-4 Weeks After Start of Treatment | 3-4 weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Number of Participants With Different Symptoms Who Had Clinical Response 6-8 Weeks After Start of Treatment | 6-8 weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Number of Participants With Different Symptoms Who Had Clinical Response 10-12 Weeks After Start of Treatment | 10-12 weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, grief, appetite disorders, and numbness) who had clinical response is presented. Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks.
Number of Participants With Clinical Response After First 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 3-4 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Clinical Response After Second 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 6-8 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Clinical Response After Third 3-4 Weeks of Treatment at 30000 IU Once Weekly Dose | 9-12 Weeks
  Clinical response to epoetin beta is characterized as an increase of hemoglobin level by >= 2 g/L against baseline with no blood transfusions within the 6 previous weeks. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors Before Receiving Treatment at 30000 IU Once Weekly | Baseline
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 3-4 Weeks After Start of Treatment at 30000 IU Once Weekly | 3-4 weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 6-8 Weeks After Start of Treatment at 30000 IU Once Weekly | 6-8 weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Different Symptoms Categorized by Lymphoproliferative Disorders and Solid Tumors 10-12 Weeks After Start of Treatment at 30000 IU Once Weekly | 10-12 Weeks
  Number of participants with different symptoms (fatigue, sleep disorders, depressed mood, lethargy, numbness, appetite disorders, and grief) is presented. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.
Number of Participants With Improvement in Symptoms Severity Categorized by Lymphoproliferative Disorders and Solid Tumors 10-12 Weeks After Start of Treatment at 30000 IU Once Weekly | 10-12 Weeks
  Number of participants with improvement in different symptoms (fatigue, depressed mood, sleep disorders, appetite disorders, lethargy, grief, and numbness) is presented. Symptoms' severity was assessed by a digital rating scale (0 to 10) of MDASI cancer participant symptom assessment questionnaire. The following severity grades were used for assessment of symptoms severity: 1) minor symptom: score 1-4; 2) moderate symptom: score 5-6; and 3) severe symptom: score 7-10. Participants who had a reduction in scores from moderate-to-severe to mild were considered improved. Results are presented for participants with lymphoproliferative disorders and solid tumors who received 30000 IU dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Russia (19):
  - Arkhangelsk
  - Barnaul
  - Belgorod
  - Ivanovo
  - Kazan'
  - Kostroma
  - Lipetsk
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Salekhard
  - Sashi
  - Surgut
  - Tver'
  - Tyumen
  - Ufa
  - Yaroslavl